CLINICAL TRIAL: NCT07306182
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetic Characteristics of SGC001 Injection in Chinese Patients With Anterior Wall ST-Segment Elevation Myocardial Infarction and Planned for Primary Percutaneous Coronary Intervention (pPCI)
Brief Title: A Research Study to Evaluate the Efficacy and Safety of SGC001 in Patients With Anterior Wall ST-Segment Elevation Myocardial Infarction
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Sungen Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SG-SGC001-201
Record Dates: First submitted 2025-12-24; First posted 2025-12-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Anterior Myocardial Infarction
MeSH Terms: conditions — Anterior Wall Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SGC001 (Experimental): Enrolled anterior STEMI patients will receive standard clinical treatment and a single dose of SGC001 on Day 1 (D1) according to their randomized dosing group. The study drug should be administered within 6 hours after the onset of acute myocardial infarction symptoms, with earlier administration preferred. The intravenous injection will be administered over 10 minutes.
  Interventions: Drug: SGC001
- Placebo (Placebo Comparator): Enrolled anterior STEMI patients will receive standard clinical treatment and a single dose of placebo on Day 1 (D1) according to their randomized dosing group. The study drug should be administered within 6 hours after the onset of acute myocardial infarction symptoms, with earlier administration preferred. The intravenous injection will be administered over 10 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SGC001 — The single dose should be administered within 6 hours after the onset of acute myocardial infarction symptoms, with earlier administration preferred. The intravenous injection should be administered over 10 minutes.
  Arms: SGC001
Drug: Placebo — The single dose should be administered within 6 hours after the onset of acute myocardial infarction symptoms, with earlier administration preferred. The intravenous injection should be administered over 10 minutes.
  Other Name
  Arms: Placebo

SUMMARY:
The research study is being done to see if SGC001 can be used to treat people scheduled to undergo percutaneous coronary intervention for Anterior ST-segment Elevation Myocardial Infarction. SGC001 might reduce the infarct size and inhibited inflammation, thereby preventing the incidence of major adverse cardiovascular events(MACE) events. Participants will either get SGC001 (active medicine) or placebo (a dummy medicine which has no effect on the body). Which treatment participants get is decided by chance. The chance of getting SGC001 or placebo is the same. The participant was administered intravenously once. SGC001 is not yet approved in any country or region in the world. It is a new medicine that doctors cannot prescribe.

ELIGIBILITY:
Inclusion Criteria:

1. 18-79 years of age (including boundary values), male or female;
2. Anterior wall STEMI: (a) history of persistent chest pain/precordial discomfort (>30 minutes); (b) upon admission, the ECG must meet the Anterior wall STEMI requirements:
3. Planned for pPCI treatment;
4. Assessed as being able to complete dosing within 6 hours of the onset of persistent chest pain/precordial discomfort symptoms;
5. The participant or their legal guardian fully understands the objectives, nature, methods, and potential adverse reactions of the study, voluntarily agrees to participate, and has signed the informed consent form (ICF).

Exclusion Criteria:

1. History of the following cardiac conditions:

   1. History of myocardial infarction, coronary revascularization (including percutaneous coronary intervention [PCI] and coronary artery bypass grafting [CABG], etc.);
   2. History of cardiopulmonary resuscitation;
   3. History of stroke;
   4. Presence of severe cardiac structural abnormalities such as aortic dissection, and ventricular aneurysm (including new-onset ventricular aneurysm);
2. Patients who have received thrombolysis;
3. Patients with a life expectancy of less than 1 year;
4. Febrile infection requiring systemic treatment within 2 weeks prior to screening;
5. Left bundle branch block (QRS duration ≥0.12 seconds. Broad R waves in leads V5 and V6, with a notch or slurring at the top, and no preceding q wave. Broad S waves or rS patterns in leads V1 and V2. T waves in leads V5 and V6 are opposite in direction to the main QRS wave);
6. Cardiogenic shock or hemodynamic instability;
7. Concomitant severe arrhythmia (including high-degree atrioventricular block, sick sinus syndrome, sustained ventricular tachycardia, etc.) or implanted cardiac pacemaker;
8. Definitive diagnosis of acute cardiac failure (Killip classification ≥ III; for details on Killip classification, see Appendix);
9. Unable to undergo cardiac magnetic resonance (CMR) imaging according to the study protocol, or known allergy to any radiocontrast agent;
10. Participation in other drug clinical trials and use of other investigational drugs within 3 months before receiving the study drug;
11. Concomitant history of the following serious diseases:

    1. Severe hepatic or renal insufficiency (e.g., requiring dialysis);
    2. Malignant tumor or history of malignant tumor;
    3. Severe autoimmune disease requiring therapeutic intervention;
12. Men and women of childbearing potential (WOCBP) who are fertile and have plans to conceive during the study period, as well as pregnant or lactating women;

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of myocardial infarction size | Day 4
  Percentage of myocardial infarction size

SECONDARY OUTCOMES:
Percentage of myocardial infarction size | Day 30, Day 90
  Percentage of myocardial infarction size
Percentage of microvascular obstruction area (MVO) | Day 4, Day 30, Day 90
  Percentage of microvascular obstruction area (MVO)
Myocardial salvage index | Day 4
  Myocardial salvage index
Left ventricular ejection fraction (LVEF) | Day 4, Day 90
  Left ventricular ejection fraction (LVEF)
Left ventricular end-systolic volume index (LVESVI) | Day 4, Day 90
  Left ventricular end-systolic volume index (LVESVI)
Left ventricular end-diastolic volume index (LVEDVI) | Day 4, Day 90
  Left ventricular end-diastolic volume index (LVEDVI)
Composite incidence of cardiovascular death | Day 90
  Composite incidence of cardiovascular death
Incidence of cardiovascular death | Day 90
  Incidence of cardiovascular death
Incidence of cardiac failure events | Day 90
  Incidence of cardiac failure events
safety endpoints | within 90 days
  Adverse events (AEs)/serious adverse events (SAEs)：physical examinations/vital signs/ECGs/laboratory tests

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will be shared when necessary